CLINICAL TRIAL: NCT00248118
Title: Neurocognitive and Affective Correlates of Tobacco Dependence in Adolescent Smokers and Efficacy and Safety of Bupropion for Treatment of Adolescent Smoking
Brief Title: Efficacy and Safety of Bupropion for Treatment of Adolescent Smoking
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI left NIH
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 999903382; 03-DA-N382
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Tobacco Dependence
Keywords: Randomized; Double-blind; Placebo-controlled
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active medication (Active Comparator): 300mg bupropion HCL
  Interventions: Drug: Bupropion
- Placebo (Placebo Comparator): Placebo pill
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Bupropion — During treatment phase, participants will take 300 mg bupropion or placebo daily.
  Other Names: Wellbutrin; Zyban

SUMMARY:
The purpose of this study is to determine: 1) the short-term clinical efficacy and safety of bupropion for helping adolescent tobacco smokers quit, and 2) The role of withdrawal symptoms in the maintenance of smoking in adolescents.

DETAILED DESCRIPTION:
This 10-week study consists of an unassisted (pretrial) acute tobacco withdrawal (AW) phase and a 7-week randomized double-blind placebo-controlled trial of bupropion (300 mg/day) for tobacco dependence. Neuropsychological examinations will be conducted at baseline, during acute withdrawal, and during treatment (incl. early withdrawal) with bupropion. We expect smoking cessation in approximately 25% of the active medication group and significant overall smoking reduction. We postulate that bupropion will also reduce the irritability, depressed mood and anxiety symptoms that typically occur during tobacco withdrawal. We expect to observe optimal cognitive performance, (i.e., attention, memory), and affective state during satiety, impairment during pre-treatment abstinence, and intermediate level cognitive performance in the abstinent active-treatment group. Because limited data are available on cognitive tasks in adolescent smokers, a non-smoking group will be included in order to establish the validity and appropriateness of our paradigm with a normative sample.

ELIGIBILITY:
Inclusion Criteria:

* More than 100 lbs
* IQ greater than 80
* General good health
* Not pregnant
* Non-Smoker: No cigarettes in last 6 months, less than 5 in lifetime
* Smokers: Smoke more than 6 cigarettes per day for at least 6 months

Exclusion Criteria:

* Cardiac, Central Nervous System (CNS) or severe psychiatric disorder
* Psychoactive medications (including nicotine replacement)
* Substance use disorder

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2005-01; Primary Completion 2007-08 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Bupropion will be safe and tolerable, increase cessation rates, and reduce smoke and nicotine exposure | 7 weeks

SECONDARY OUTCOMES:
Reduction of smoking-related urges and cravings. | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric T. Moolchan, M.D., Principal Investigator — National Institute on Drug Abuse, Intramural Research Program
Locations (1):
- Teen Tobacco Addiction Research Clinic, NIDA Intramural Research Program, Baltimore, Maryland, United States